CLINICAL TRIAL: NCT00829361
Title: Stroke Telemedicine for Arizona Rural Residents Trial
Acronym: STARR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona Department of Health Services (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-005156
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Stroke; Cerebral Infarction; Vascular Diseases; Brain Ischemia; Brain Infarction; Brain Diseases; Cerebrovascular Disorders
Keywords: Telemedicine; Acute stroke; Rural; thrombosis; consultation; Stroke; Cerebral Infarction; Vascular diseases; brain ischemia; brain infarction; brain diseases; cerebrovascular disorders
MeSH Terms: conditions — Stroke; Cerebral Infarction; Vascular Diseases; Brain Ischemia; Brain Infarction; Brain Diseases; Cerebrovascular Disorders; Thrombosis | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Telemedicine (Other)
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — Two way site independent audio/video telemedicine system with DICOM.

SUMMARY:
The STARR network registry consists of a 4 spoke 1 hub system. Which will consist of prospective collection, recording, and regular analysis of telestroke patient consultation and care data for the purpose of quality measure assessment and improvement and benchmarking against other national and international telestroke programs.

DETAILED DESCRIPTION:
Background:

Acute stroke resources and care are deficient in Arizona's rural communities. Stroke telemedicine is a proven modality for overcoming the deficiency. Stroke telemedicine allows a telephonic consultation and/or two-way audio video consultation between a stroke neurologist and a stroke patient at a remotely located emergency department. University of California San Diego Stroke Center has completed an NIH funded randomized controlled trial, STRokE DOC, comparing telephonic consultations to video consultations. In that trial, video telemedicine consultations resulted in more accurate decision making compared with telephone consultations. The video telemedicine consultative modality provides the rural stroke patient with the opportunity to receive expert stroke care, interpretation of neuroimaging, determination of appropriate acute therapy, and recommendations regarding need for transfer to a higher level of care. Mayo Clinic Arizona is currently completing a state funded feasibility trial, STRokE DOC Arizona (06-005731), as a preliminary step toward establishing a state wide stroke telemedicine network, STARR. The STARR network plan should include the prospective collection, recording, and regular analysis of telestroke patient consultation data for the purpose of quality measure assessment and improvement.

Objective:

The objective of this research is to establish a system for the prospective collection, recording, and regular analysis of telestroke patient consultation and care data for the purpose of quality measure assessment and improvement and benchmarking against other national and international telestroke programs.

Methods:

The STARR network consists of a primary stroke center hub (Mayo Clinic Hospital) that serves multiple spoke hospitals in remote and rural regions of the state (e.g. Kingman and Yuma Regional Medical Centers, La Paz Regional Hospital and Copper Queen Community Hospital). Mayo Clinic vascular neurologists, who have licenses and privileges to practice teleneurology at spoke hospitals in the state, participate in a 24/7 Mayo Clinic telestroke hotline. When an acute stroke patient presents to a STARR network participating spoke hospital emergency department, a stroke alert is activated and the hotline is phoned. An on-call vascular neurologist receives the pager notification and communicates with the referring emergency physician. The telestroke consultation will begin by telephone and will be supplemented by audio-video telemedicine communication and teleradiology. The patient is registered at Mayo Clinic and a registration number is generated by the house supervisor. Emergency neurology care is rendered. Every participating spoke hospital emergency physician is already a sub-investigator in telestroke research and has completed HSRP training and certification. The Mayo Clinic IRB has served as the central IRB of record for state funded Mayo Clinic telestroke research. The patient or legal designate will be approached by either the spoke emergency physician investigator and/or the hub neurologist investigator (via telemedicine camera) for consent to proceed with telestroke consultation, and to acquire, store, and analyze data concerning the acute stroke care and outcome of the patient. Data sources will include the Mayo Clinic electronic transcribed telestroke consultation note, the emergency department nursing and physician records, the admission consultation and diagnostic tests records, hospital discharge note, and the content of a brief 90 day follow-up phone call by the research coordinator to patient and/or family member. The licensed neurologists already have authorization to access patient spoke hospital records as part of their clinical privileges, but the designated Mayo Clinic research coordinator will have the responsibility to extract data from the sources and enter it into the registry. The STARR registry data elements will be exactly the same as the established and familiar data elements for the STRokE DOC Arizona trial, for the purposes of continuity. Mayo Clinic Arizona research biostatistics group will develop the electronic data manager and conduct and report analyses monthly to the telestroke research group.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Rural Emergency Department within 12 hours of acute stroke symptom onset.
* Written informed consent.

Exclusion Criteria:

* Unlikely to complete study through 90-day follow-up.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To assess the numbers of patients who receive thrombolytics and the time to treatment in patients evaluated by telemedicine | 90 days

SECONDARY OUTCOMES:
To assess the functional outcomes of acute stroke subjects by Barthel index and Modified Rankin Scale | 90 days
To assess the rate of intracranial hemorrhage post thrombolysis | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Bart M. Demerschalk, M.D., Principal Investigator — Mayo Clinic; Bentley J. Bobrow, M.D., Principal Investigator — Mayo Clinic; Dwight D Channer, MS, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic Hospital, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Demaerschalk BM, Aguilar MI, Ingall TJ, Dodick DW, Vargas BB, Channer DD, Boyd EL, Kiernan TEJ, Fitz-Patrick DG, Collins JG, Hentz JG, Noble BN, Wu Q, Brazdys K, Bobrow BJ. Stroke Telemedicine for Arizona Rural Residents, the Legacy Telestroke Study. Telemed Rep. 2022 Mar 14;3(1):67-78. doi: 10.1089/tmr.2022.0002. eCollection 2022. PMID 35720454
- [Derived] Demaerschalk BM, Vargas JE, Channer DD, Noble BN, Kiernan TE, Gleason EA, Vargas BB, Ingall TJ, Aguilar MI, Dodick DW, Bobrow BJ. Smartphone teleradiology application is successfully incorporated into a telestroke network environment. Stroke. 2012 Nov;43(11):3098-101. doi: 10.1161/STROKEAHA.112.669325. Epub 2012 Sep 11. PMID 22968466
- [Derived] Capampangan DJ, Wellik KE, Bobrow BJ, Aguilar MI, Ingall TJ, Kiernan TE, Wingerchuk DM, Demaerschalk BM. Telemedicine versus telephone for remote emergency stroke consultations: a critically appraised topic. Neurologist. 2009 May;15(3):163-6. doi: 10.1097/NRL.0b013e3181a4b79c. PMID 19430275